CLINICAL TRIAL: NCT04287725
Title: Additional Effects Of The Association Of The Photobiomodulation Therapy (904 Nm) With Exercise In Participants With Chronic Non-Specific Low Back Pain In The Long Term
Brief Title: Effects of Laser Therapy and Exercise in Participants With Chronic Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federal University of the Valleys of Jequitinhonha and Mucuri (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18022020
Record Dates: First submitted 2020-02-18; First posted 2020-02-27 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Low Back Pain (LBP)
MeSH Terms: conditions — Low Back Pain | interventions — Exercise Therapy; Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercise + active Photobiomodulation therapy (PBMT) (Experimental): Exercise protocol: The program will consist of individual sessions of progressive and submaximal exercises with aerobic training on a treadmill and spine strengthening exercise.
  Photobiomodulation therapy: will be performed using the active super pulsed laser (904nm).
  Interventions: Device: exercise + photobiomodulation therapy
- exercise + placebo Photobiomodulation therapy (PBMT) (Placebo Comparator): Exercise protocol: The program will consist of individual sessions of progressive and submaximal exercises with aerobic training on a treadmill and spine strengthening exercise.
  Photobiomodulation therapy: will be performed using the placebo super pulsed laser (904nm).
  Interventions: Device: exercise + photobiomodulation therapy

INTERVENTIONS:
Device: exercise + photobiomodulation therapy — Treatment sessions will be provided twice a week for 6 weeks (totaling 12 sessions) with participants receiving either placebo or active PBMT + exercise protocol.

SUMMARY:
The objective of this clinical trial is to evaluate the additional effects of Laser Therapy in participants with chronic non-specific low back pain in the short and long term.

DETAILED DESCRIPTION:
The objective of this clinical trial is to evaluate the additional effects of Photobiomodulation Therapy in participants with chronic non-specifc low back pain in the short and long term.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-specific chronic LBP, defined as pain or discomfort between the costal margins and inferior gluteal folds with or without referred pain to the lower limbs;
* Persistent LBP for at least 3 months;
* Low back pain of intensity reported 3 or higher by the Visual Analogue Scale (VAS), at least once in the previous 7 days;
* Aged between 18 and 65 years;
* Both genders.

Exclusion Criteria:

* Patients with severe skin diseases (eg, skin cancer, erysipelas, severe eczema, severe dermatitis, severe psoriasis and severe hives lupus);
* Participants with known or suspected serious spinal pathology (e.g., fractures, tumors, inflammatory, rheumatologic disorders, or infective diseases of the spine);
* Nerve root compromise;
* History of previous spinal surgery (even in a segment other than the lumbar spine) or scheduled surgery;
* Pain due to or associated with pregnancy or structural deformity (for example, scoliosis);
* Pregnancy;
* Comorbid health conditions that could prevent active participation in the exercise programs such as high blood pressure, pregnancy, or cardio-respiratory illnesses;
* Having answered "yes" to any of the questions in the Physical Activity Readiness Questionnaire (PAR-Q);
* Be treated with PBMT;
* Being under physiotherapeutic treatment or perform physical exercise;
* Who are using NSAID or start it during the trial;
* Who have inability to tolerate the proposed experimental procedures (such as tests of mobility and strength of the lumbar muscles).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2021-06-02 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change Of Pain intensity at post-intervention | Baseline; Immediately after the last intervention
  Measured by the Visual Analogue Scale (VAS). The VAS evaluates pain intensity levels perceived by the patient on an 11-point scale ranging from 0 to 10, with 0 being 'no pain' and 10 'the worst possible pain'.
Change Of Pain intensity at 3 months post-intervention | Baseline; 3 months after the last intervention
  Measured by the Visual Analogue Scale (VAS). The VAS evaluates pain intensity levels perceived by the patient on an 11-point scale ranging from 0 to 10, with 0 being 'no pain' and 10 'the worst possible pain'.
Change of Disability associated with low back pain at post-intervention | Baseline; Immediately after the last intervention
  Measured by the Roland-Morris Disability Questionnaire. The questionnaire consists of 24 items that describe situations that patients may have difficulty performing on a daily basis due to LBP. The greater the number of affirmative answers is, the higher the level of functional disability associated with LBP.
Change of Disability associated with low back pain at 3 months post-intervention | Baseline; 3 months after the last intervention
  Measured by the Roland-Morris Disability Questionnaire. The questionnaire consists of 24 items that describe situations that patients may have difficulty performing on a daily basis due to LBP. The greater the number of affirmative answers is, the higher the level of functional disability associated with LBP.

SECONDARY OUTCOMES:
Change Of Pain intensity at 12 months post-intervention | Baseline; 12 months after the last intervention
  Measured by the Visual Analogue Scale (VAS). The VAS evaluates pain intensity levels perceived by the patient on an 11-point scale ranging from 0 to 10, with 0 being 'no pain' and 10 'the worst possible pain'.
Change of Disability associated with low back pain at 12 months post-intervention | Baseline; 12 months after the last intervention
  Measured by the Roland-Morris Disability Questionnaire. The questionnaire consists of 24 items that describe situations that patients may have difficulty performing on a daily basis due to LBP. The greater the number of affirmative answers is, the higher the level of functional disability associated with LBP.
Changes os Mental health | Baseline; Immediately after the last intervention; 3 and 12 months after the last intervention
  Measured by the reduced version of the Anxiety, Depression and Stress Scale-21. It is a self-report instrument composed of three subscales with seven items each, to assess depression, anxiety and stress in the previous week. The variations in scores correspond to symptom levels, which vary between "normal" and "very severe".
Changes of Disability associated with low back pain | Baseline; Immediately after the last intervention; 3 and 12 months after the last intervention
  Measured by the Oswestry Low Back Pain Disability Questionnaire. The scale consists of 10 questions with six alternatives, the value of which ranges from 0 to 5. It is classified into: minimum disability (0 - 20%), moderate disability (21- 40%), severe disability (41 - 60%) , a patient who is disabled (61 - 80%), and an individual restricted to bed (81 - 100%).
Changes of Mobility of the lumbar and sacral segments | Baseline; Immediately after the last intervention; 3 and 12 months after the last intervention
  Measured by the modified Schober test
Changes of Strength of the trunk extensor muscle | Baseline; Immediately after the last intervention; 3 and 12 months after the last intervention
  Measured by the Sorensen Test

CONTACTS AND LOCATIONS:
Overall Officials: Flávia Santos, Principal Investigator — Federal University of the Valleys of Jequitinhonha and Mucuri

IPD SHARING:
Plan to Share IPD: No